CLINICAL TRIAL: NCT03516344
Title: Effect of Osteopathic Manipulations on Portal Venous Flow: Randomized Clinical Trial
Brief Title: Effect of Osteopathic Manipulations on Portal Venous Flow
Acronym: ECOPORTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Antonio de Nebrija (Other)
Responsible Party: Principal Investigator, José Ríos-Díaz, Principal Investigator, Universidad Antonio de Nebrija
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Eco_Porta
Record Dates: First submitted 2018-03-23; First posted 2018-05-04 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Breathing Exercises; Manipulation, Osteopathic; Physical Therapy; Ultrasonography; Portal Vein
Keywords: Breathing Exercises; Manipulation, Osteopathic; Quantitative Ultrasonography; Therapy, Soft Tissue; Portal Vein; Venous flow
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): Subjects will remain at rest in supine position for one minute.
- Iliac psoas muscle (Experimental): In supine position with a high-density foam cushion under the subject's feet, they will be asked to make a push in the caudal direction, against the cushion, alternating between both feet with their knees stretched out, for one minute
  Interventions: Procedure: Liver pumping and Spinal manipulation
- Diaphragmatic Breathing (Experimental): Subjects perform five cycles of diaphragmatic breathing in the supine position.
  Interventions: Procedure: Liver pumping and Spinal manipulation
- Liver pumping (Experimental): A technique of hepatic supine pumping is performed by simultaneous compression in the right hypochondrium and epigastrium, in the opposite direction, during the inspiratory phase, stopping during the expiratory phase and repeating the maneuver for five respiratory cycles.
  Interventions: Procedure: Liver pumping and Spinal manipulation
- Spinal manipulation (Experimental): A semi-direct vertebral manipulation, type Dog Technique in extension, will be performed on level D8
  Interventions: Procedure: Liver pumping and Spinal manipulation

INTERVENTIONS:
Procedure: Liver pumping and Spinal manipulation — Interventions are described in group descriptions
  Other Names: Vertebral manipulation; Soft tissues mobilization
  Arms: Diaphragmatic Breathing; Iliac psoas muscle; Liver pumping; Spinal manipulation

SUMMARY:
Since osteopathy it is considered that the alterations in the mobility of the different structures of the organism could cause a decrease in the blood circulation of the tissue causing a functional disorder and, with time, the appearance of a disease.

In visceral osteopathy, the treatment of liver dysfunctions it is important due to their interrelation with the functioning of the rest of the abdominal and pelvic viscera and, especially, through the hepatic portal system. However, there are few studies showing whether a manual therapeutic intervention can affect the mobility, function or vascularization of a viscera.

Ultrasonography is an appropriate tool for validating some of these intervention procedures given their safety, repeatability, autonomy and the low cost of the procedures and technical equipment which, in a non-invasive manner, will allow the effects of the different therapeutic interventions to be verified.

Hypothesis:

1. Vertebral manipulations and pumping of the liver improve the flow of the portal vein in front of the diaphragmatic breathing and the contraction of the psoas iliac muscle.
2. The accuracy of ultrasound to assess venous flow may be useful as an outcome measure.

Objectives: To describe the immediate changes of different manipulative interventions on portal vein flow in healthy women and to obtain baseline measurements for future research.

Sample description: Pilot randomized controlled clinical trial with a sample of 50 healthy adult women recruited intentionally sampled that will be pseudo-randomly forcing equality of groups: control, chest manipulation, liver manipulation, abdominal breathing and iliac psoas muscle contraction.

The minimum size required has been calculated using the program G*Power 3.1.3 for Windows (University Kiel, Germany, 2008) based on an effect size of 0.5, type I error of 5%,type II error of 10% and an effect size of f=0.45.

DETAILED DESCRIPTION:
The non-invasive intervention procedure in each of the groups is as follows:

1. Control group (CG): Subjects will remain at rest in supine position for one minute.
2. Thoracic manipulation group (GMT): A semi-direct vertebral manipulation will be performed, type Dog Technique in extension, above level D8.
3. Liver manipulation group (HMG): A supine hepatic pumping technique will be performed, performing simultaneous compression in the right hypochondrium and epigastrium, in the opposite direction, during the inspiratory phase, stopping during the expiratory phase and repeating the maneuver for five respiratory cycles.
4. Abdominal breathing group (GRA): Subjects will be asked to perform five cycles of diaphragmatic breathing in the supine position.
5. Psoas exercise group (GPS): In the supine position with a high density foam cushion under the feet of the subject, it will be asked to make a push in the caudal direction, against the cushion, alternating between both feet with the knees stretched, for one minute.

After informed consent and recording of personal data, participants will be placed in a constant and regulated temperature room where they will be placed in supine position for 5 minutes for cardiocirculatory normalization, at least 2 hours after the last meal. The room where the explorations will be carried out is conditioned to keep the ambient temperature constant.

The study will be carried out with independent recruitment and triple blinding: the patient will not know the intervention group, the sonographer will not know the technique applied to the patients, the researcher responsible for recording the flows and diameters and the temperature will also be masked and the data analyst will be masked during the statistical analysis process.

For statistical analysis, a descriptive analysis using means and standard deviations will be performed, as well as ranges and quartiles for quantitative measurements. Qualitative variables shall be summarised by counts and frequencies. The assumption of normality (Shapiro-Wilks test) and equality of variances (Levene's test) prior to the analysis of variance (ANOVA) will be checked for repeated measurements in which the intra-unit factors (three time measurements) will be the dependent variables (velocity, diameter and temperature) and the inter-subject factor, the study group. If it is not possible to assume the application assumptions, the corresponding non-parametric tests will be chosen. Pair comparisons were made with the Dunn-Bonferroni correction for type I erro and the age and BMI variables were entered into the model as covariates to estimate their possible effect on the dependent variables. The percentages of change from the baseline values in the intra-group comparison and from the control group in the intergroup comparison shall be calculated. The effect size will be estimated with the Hedges g statistic.

The significance level will be set to p<0.05 and calculations will be performed with SPSS 19.0

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* No history of abdominal surgery or liver disease

Exclusion Criteria:

* Fear or apprehension of techniques

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Flow velocity of the portal vein | Pre-intervention, immediately post-intervention and 5-minutes-post-intervention
  In cm/s, FV is obtained from ultrasound scans (General Electric LogiqE ultrasound scanner model with the 4C-RS convex probe with a working frequency of 2-5 MHz.).
  All image optimization parameters remained constant for all patients and scans. The records will be made by a researcher with 15 years of ultrasound experience.
Diameter of the portal vein | Pre-intervention, immediately post-intervention and 5-minutes-post-intervention
  In mm, DIA is obtained from ultrasound scans (General Electric LogiqE ultrasound scanner model with the 4C-RS convex probe with a working frequency of 2-5 MHz.).
  All image optimization parameters remained constant for all patients and scans. The records will be made by a researcher with 15 years of ultrasound experience.

SECONDARY OUTCOMES:
Temperature of D7-D8 dermatome | Pre-intervention, immediately post-intervention and 5-minutes-post-intervention
  The temperature of the dermatome D7-D8, in relation metameric to the liver, is recorded at the xiphoid process level with an infrared thermometer (ºC)

CONTACTS AND LOCATIONS:
Locations (1):
- José Ríos-Diaz, Madrid, Spain

REFERENCES:
- [Background] Allan PL, Ph.D WNM, Pozniak MA, Dubbins PA. Ecografía doppler clínica. Elsevier España; 2008.
- [Background] Allan PLP, Baxter GM, Weston M. Clinical Ultrasound. 3rd ed. Philadelphia: Churchill Livingstone Elsevier, 2011
- [Background] Baert AL, Brady LW, Heilmann HP, Molls M, Sartor K. Duplex and color doppler imaging of the venous system. Springer; 2014.
- [Background] Harris W, Wagnon RJ. The effects of chiropractic adjustments on distal skin temperature. J Manipulative Physiol Ther. 1987 Apr;10(2):57-60. PMID 3585197
- [Background] Hebgen E. Osteopatía Visceral. Fundamentos y técnicas. 2ª edición ed. Madrid: McGraw-Hill. Interamericana; 2005
- [Background] Korr IM. Bases fisiologicas de la osteopatía. 1ª ed.: Mandala; 2004
- [Background] Martínez-Payá JJ, de-Groot-Ferrando A, Ríos-Díaz J, del-Baño-Aledo ME. Sonoanatomy of the musculoskeletal system. En: Valera F, Minaya F, editores. Advanced Techniques in Musculoskeletal Medicine & Physiotherapy. Edinburgh: Churchill Livingstone; 2016. p.147-70.
- [Background] Resende C, Lessa A, Goldenberg RCS. Ultrasonic Imaging in Liver Disease: From Bench to Bedside. Rijeka, Croatia: INTECH Open Access Publisher; 2011.p.127-56.
- [Background] Ricard F. Tratado de osteopatía visceral y medicina interna. Tomo 2: Sistema digestivo. 1ª edición ed. Madrid: Editorial Médica Panamericana; 2008
- [Background] Welch A, Boone R. Sympathetic and parasympathetic responses to specific diversified adjustments to chiropractic vertebral subluxations of the cervical and thoracic spine. J Chiropr Med. 2008 Sep;7(3):86-93. doi: 10.1016/j.jcm.2008.04.001. PMID 19646369